CLINICAL TRIAL: NCT04238767
Title: Observational Assessment of the Nation-wide Roll-out of Dolutegravir in Lesotho
Brief Title: Dolutegravir in Real Life in Lesotho
Acronym: DO-REAL
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: SolidarMed (Other); Ministry of Health, Lesotho (Other Government); District Health Management Team of Butha-Buthe, Lesotho (Other); District Health Management Team of Mokhotlong, Lesotho (Other); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: P001-19-1.2
Record Dates: First submitted 2019-11-14; First posted 2020-01-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-10

CONDITIONS: HIV-1-infection
Keywords: HIV-1; AIDS; dolutegravir; antiretroviral therapy; Lesotho; sub-Saharan Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1-positive individuals: HIV-1-positive individuals eligible to receive a DTG-based ART regimen at enrolment.
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Eligibility to receive DTG-based ART at enrolment (i.e., initiation or offer to initiate DTG-based ART)

SUMMARY:
DO-REAL is an observational cohort study assessing the large-scale roll-out of the antiretroviral drug dolutegravir (DTG) in Lesotho.

DTG has been shown to have low side-effects and superior treatment outcomes for people living with HIV-1 when compared to other antiretroviral drugs currently in use in low-income countries. The use of DTG in first-line antiretroviral therapy (ART) regimens was recommended by the World Health Organisation in 2018 and adopted by the Ministry of Health in Lesotho in 2019. While DTG-based ART regimens have led to promising health outcomes in high-income and clinical trial settings, certain concerns remain regarding the risk of ART-experienced patients transitioning to a DTG-based ART regimen being placed on a functional monotherapy (increasing the otherwise low risk of viral resistance to DTG) as well as side-effects including psychological symptoms and weight gain.

Thus, the DO-REAL study intends to address these concerns and provide data on health outcomes of HIV patients on DTG in a "real-life" high-prevalence setting.

DETAILED DESCRIPTION:
SUMMARY: DO-REAL is an observational cohort study assessing the large-scale roll-out of the antiretroviral drug dolutegravir (DTG) in Lesotho.

BACKGROUND: DTG is a second-generation integrase strand transfer inhibitor with low side-effects and superior treatment outcomes for people living with HIV-1 when compared to other antiretroviral drugs currently in use in low-income countries. Though some cases have been described, HIV-1 resistance to DTG is rare in clinical settings when DTG is used as part of a combination therapy. The use of DTG in first-line antiretroviral therapy (ART) regimens was recommended by the World Health Organisation in 2018 and was adopted by the Ministry of Health in Lesotho in 2019. DTG now forms part of the recommended first-line therapy for many ART-naïve patients in Lesotho. In addition, many patients on a non-DTG-based first-line ART regimen will be transitioned to a DTG-based regimen.

OBJECTIVES: Despite the positive health outcomes observed in patients receiving DTG-based ART in high-income countries and in clinical trial settings, there is little data on virologic outcomes of patients on DTG during large-scale implementation in low- and lower middle-income countries. Concerns remain regarding the risk that some patients transitioning to a DTG-based regimen will be placed on a functional monotherapy. Furthermore, there are concerns as to psychological side-effects and observed weight gain. This observational study aims to assess the virologic outcomes (viral suppression rates as well as potential drug resistance) as well as side-effects of people living with HIV-1 and transitioning to a DTG-based ART regimen in Lesotho.

DO-REAL has two major objectives:

* To assess virologic outcomes after the programmatic shift to DTG-based regimens.
* To assess psychological and somatic wellbeing in patients before and after the programmatic shift to DTG-based regimens.

METHODS: DO-REAL is a cohort study enrolling people living with HIV who are initiating or are eligible (according to national guidelines and the local implementation thereof) to initiate a DTG-based antiretroviral therapy (ART) regimen. The study will take place at three hospitals in two districts (Butha-Buthe, Mokhotlong) in Lesotho, and aims to enrol over 2000 participants. Viral loads will be measured on the day of initiating a DTG-based regimen (or on the day this was offered), as well as four, 12 and 24 months thereafter. In a post-hoc analysis, samples will be tested for drug resistance in samples where the viral load permits (approx. ≥100 c/mL). A subset of participants will complete screenings for depression, general health, and HIV-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-positive
* Initiating or eligible to initiate (offered to initiate) a DTG-based ART regimen
* Informed written consent (and assent, if applicable) provided

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be enrolled at two government hospitals and one missionary hospital in two districts (Butha-Buthe and Mokhotlong) in Lesotho.
Sampling Method: Non-Probability Sample
Enrollment: 1433 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Virologic outcomes after programmatic transition to DTG-containing regimens | 4 months after initiation of a DTG-containing regimen
  Viral load
Quality of life screening score (change from baseline) | Change between time of initiation of a DTG-containing ART regimen and 4 months thereafter
  12-Item Short Form Health Survey (SF-12; 12-item index in which questions are scored and weighted into 2 subscales, physical health and mental health; scores can range from 0-100 with higher scores indicating higher physical or mental health)
Depression screening score (change from baseline) | Change between time of initiation of a DTG-containing ART regimen and 4 months thereafter
  Patient Health Questionnaire-9 (PHQ-9; 9-item index with each item scored 0-3, providing a 0-27 severity score with a higher score indicating higher severity)
HIV symptom screening score (change from baseline) | Change between time of initiation of a DTG-containing ART regimen and 4 months thereafter
  Modified HIV Symptom Index (21-item index with each item scored 0-4, providing a 0-84 severity score with a higher score indicating higher severity)

SECONDARY OUTCOMES:
Virologic status at programmatic transition to DTG-containing regimens | On day of initiation of a DTG-containing regimen
  Viral load (post-hoc analysis)
Viral drug resistance at programmatic transition to DTG-containing regimens | On day of initiation of a DTG-containing ART regimen
  HIV-1 drug resistance (assessed by Sanger sequencing) in the case of an unsuppressed viral load (post-hoc analysis)
Weight (change from baseline) | On day of initiation of a DTG-containing ART regimen and 4, 12 and 24 months thereafter
  Change from time of enrolment; median and interquartile range; in kg
Reasons for discontinuation of a DTG-containing regimen | Up to 24 months after enrolment
  Reasons for discontinuing a DTG-containing regimen as noted in medical records, where applicable
Long-term virologic outcomes after programmatic transition to DTG-containing regimens | 12 and 24 months after initiation of a DTG-containing regimen
  Viral load
Viral drug resistance after programmatic transition to DTG-containing regimens | 4, 12 and 24 months after initiation of a DTG-containing regimen
  HIV-1 drug resistance (assessed by Sanger sequencing) in the case of an unsuppressed viral load

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus D Labhardt, MD, MIH, Study Chair — Swiss Tropical & Public Health Institute; Thomas Klimkait, PhD, Study Director — University of Basel; Josephine Muhairwe, MD, MPH, Study Director — SolidarMed; Jennifer A Brown, MSc, MAS D&C, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- Lesotho (2):
  - Butha-Buthe Government Hospital, Butha-Buthe
  - Seboche Mission Hospital, Butha-Buthe

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized dataset for the published manuscripts "Viral suppression after transition from nonnucleoside reverse transcriptase inhibitor- to dolutegravir-based antiretroviral therapy: A prospective cohort study in Lesotho (DO-REAL study)" and "Dolutegravir in Real Life: self-reported mental and physical health outcomes after transitioning from efavirenz- to dolutegravir-based antiretroviral therapy in a prospective cohort study in Lesotho" are publicly available on Zenodo:
  https://zenodo.org/record/5948369 https://zenodo.org/record/6654462

REFERENCES:
- [Result] Brown JA, Nsakala BL, Mokhele K, Rakuoane I, Muhairwe J, Urda L, Amstutz A, Tschumi N, Klimkait T, Labhardt ND. Viral suppression after transition from nonnucleoside reverse transcriptase inhibitor- to dolutegravir-based antiretroviral therapy: A prospective cohort study in Lesotho (DO-REAL study). HIV Med. 2022 Mar;23(3):287-293. doi: 10.1111/hiv.13189. Epub 2021 Oct 10. PMID 34632682
- [Result] Brown JA, Nsakala BL, Mokhele K, Rakuoane I, Muhairwe J, Glass TR, Amstutz A, Tschumi N, Belus JM, Klimkait T, Labhardt ND. Dolutegravir in real life: Self-reported mental and physical health outcomes after transitioning from efavirenz- to dolutegravir-based antiretroviral therapy in a prospective cohort study in Lesotho. HIV Med. 2023 Feb;24(2):153-162. doi: 10.1111/hiv.13352. Epub 2022 Jun 22. PMID 35730213
- Available data/document: Individual Participant Data Set: 10.5281/zenodo.6654462 — https://zenodo.org/record/6654462 — Dataset relating to: Brown JA, Nsakala BL, Mokhele K, et al. Dolutegravir in real life: Self-reported mental and physical health outcomes after transitioning from efavirenz- to dolutegravir-based antiretroviral therapy in a prospective cohort study in Lesotho. HIV Med. Published online June 22, 2022. doi:10.1111/hiv.13352
- Available data/document: Individual Participant Data Set — https://zenodo.org/record/5948369 — Dataset relating to: Brown JA, Nsakala BL, Mokhele K, et al. Viral suppression after transition from nonnucleoside reverse transcriptase inhibitor- to dolutegravir-based antiretroviral therapy: A prospective cohort study in Lesotho (DO-REAL study). HIV Med. 2022;23(3):287-293. doi:10.1111/hiv.13189